CLINICAL TRIAL: NCT01127529
Title: Ceprotin Treatment Registry
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: UDC Rare Bleeding and Clotting Disorders Working Group (RBDWG) (Unknown); American Thrombosis and Hemostasis Network (Network)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 400701
Record Dates: First submitted 2010-04-16; First posted 2010-05-21 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Protein C Deficiency
MeSH Terms: conditions — Protein C Deficiency | interventions — Protein C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with severe congenital protein C deficiency: Registry subjects will be identified by working with Hemophilia Treatment Centers and Thrombosis Centers known to have subjects with severe congenital protein C deficiency, as well as by working with centers that use Ceprotin in emergency care situations.
  Interventions: Biological: Protein C Concentrate (Human)

INTERVENTIONS:
Biological: Protein C Concentrate (Human) — Commercially available Ceprotin will be prescribed, obtained and administered by the investigator according to local standard of care.
  Other Names: Ceprotin

SUMMARY:
The overall objective is to collect and assess data on the treatment, safety, and treatment outcomes of subjects prescribed, receiving and participating in the Ceprotin treatment registry.

ELIGIBILITY:
Inclusion Criteria:

Participants for whom CEPROTIN therapy has been indicated and meeting the following criteria may be enrolled in this study:

* Signed and dated informed consent from either the participant or the participant's legally authorized representative prior to enrollment, as applicable
* Males and females of any age, including neonates, children, adolescents and adults
* Participant who received CEPROTIN or is initiating/receiving CEPROTIN treatment

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Registry participants will be identified by working with Hemophilia Treatment Centers and Thrombosis Centers known to have participants with severe congenital Protein C deficiency, as well as by working with centers that use CEPROTIN in emergency care situations.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2010-06-23 (Actual); Primary Completion 2015-06-22 (Actual); Study Completion 2015-06-22 (Actual)

PRIMARY OUTCOMES:
Medical diagnoses associated with Ceprotin treatment | 2 to 5 years, or until the Registry is terminated
Ceprotin treatment regimens | 2 to 5 years, or until the Registry is terminated
Safety information based on all serious adverse events (SAEs), related SAEs and related non-serious adverse events (AEs) | 2 to 5 years, or until the Registry is terminated

SECONDARY OUTCOMES:
Treatment outcomes categorized by medical diagnosis | 2 to 5 years, or until the Registry is terminated
  Evidence of halting or reversal of coagulopathy or thrombosis, end-organ damage, limb sparing, Length of Hospital Stay (LOS), and mortality
CEPROTIN use and treatment outcomes in pregnancy, labor and delivery, surgery and invasive procedures, different age groups, and, in the presence of pre-existing renal and/or hepatic dysfunction | 2 to 5 years, or until the Registry is terminated

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (28):
- United States (12):
  - Phoenix, Arizona
  - Orange, California
  - Aurora, Colorado
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - Lebanon, New Hampshire
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Fort Worth, Texas
  - Houston, Texas
- Austria (2):
  - Innsbruck
  - Vienna
- Germany (6):
  - Bonn
  - Frankfurt
  - Hanover
  - Heidelberg
  - Magdeburg
  - Magstadt
- Italy (4):
  - Milan
  - Palermo
  - Rome
  - Vicenza
- Nijmegen, Netherlands
- United Kingdom (3):
  - Bradford
  - London
  - Manchester

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fc84db2bf003ab460cc